CLINICAL TRIAL: NCT06138002
Title: Randomized Clinical Investigation to Assess Preliminary Clinical Performance, Effectiveness and Safety of the LumbaCure® (prototype C190070.01) Medical Device When Used in Patients Suffering from Chronic Low Back Pain
Brief Title: Clinical Investigation to Assess the Clinical Performance of the LumbaCure® Intervention on Chronic Low Back Pain Patients.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Design change
Sponsor: Odix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIV-23-05-043012
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Intervention arm (Experimental): The LumbaCure® is a robotic system which provide active, specific and controlled mobilization of the low back. The device is to be used by the Physiotherapist at the rehabilitation centre. The duration of a session for the patient is 15 minutes.
  Patients follow a serie of 12 consecutive LumbaCure® sessions at a frequency of 3 sessions / week for 4 weeks.
  Interventions: Device: LumbaCure®
- Control Intervention arm (Active Comparator): A set of core stability exercises/active qualitative mobilization has been defined with principal investigator according to the standard of care at Investigator site. At each session, 5 exercises will be selected by the investigator depending on the evolution and pathology of the patient. Five minutes of warm-up will be performed before starting the exercises session.
  The program will last 15 to 30 min depending on the time required for the patient to complete the prescribed exercises.
  Patients follow a serie of 12 consecutive physical exercises sessions at a frequency of 3 sessions / week for 4 weeks.
  Interventions: Procedure: Physical Exercises supervised by the physiotherapist

INTERVENTIONS:
Device: LumbaCure® — LumbaCure®is a robotic system that systematically moves the spine of affected patients with a complex proprietary algorithm.
  Arms: Test Intervention arm
Procedure: Physical Exercises supervised by the physiotherapist — A set of core stability/active qualitative mobilization exercises have been defined, corresponding to standard exercises proposed in center rehabilitation program
  Arms: Control Intervention arm

SUMMARY:
Low Back Pain (LBP) is one of the common causes of morbidity worldwide, with a one-month prevalence of 23.3 %. Number of people with LBP reached 577 million people in 2020. LBP has been the leading cause of years lived with disability from 1990 to 2017. The highest incidence of LBP is in people in their third decade of age. LBP is a complex disease difficult to treat as most of these cases (80 - 90 %) are classified as non-specific meaning that the pain cannot be attributed to any specific injury or pathology.

Until now exercise therapy is commonly used as the treatment of choice in the revalidation program of LBP. The aim of physical treatment is to improve function and prevent disability from getting worse.

LumbaCure® is a robotic system driven by a proprietary movement algorithm to induce a specific and controlled mobilization of the hips and the low back in patient requiring treatment by physical exercises due to orthopedic disorder, especially low back pain.

The investigation include an intervention period of 4 weeks The main objective is to compare the impact on disability (Oswestry disability Index) and movement performance of the interventions (LumbaCure® vs physical exercises supervised by the physiotherapist) in two parallel groups of patients suffering from chronic low back pain.

The investigation includes an intervention period of 4 weeks and a follow-up period of 6 months (post intervention period).

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific LBP (without red flag)
* Patient did not increase, on a long-term basis, his/her regular physical activity in the past 2 months.
* LBP is the principal musculoskeletal condition
* Aged between 18 and 65 years old
* Able to read and understand questionnaires and communicate with the physiotherapist.
* Average Back Pain intensity over the last week above 2, assessed on Numerical Pain Rating Scale from 0 to 10 anchored with "no pain" at 0 and "worst pain imaginable " at 10.
* ODI score > 20

Exclusion Criteria:

* Suspected or confirmed serious pathology (i.e infection, fracture, cancer, inflammatory arthritis, ….)
* Radicular pain
* Radiculopathy
* Cognitive impairment that precludes participant from consenting, completing investigation questionnaires or complying with recommendations
* Previous spine surgery in the last 3 months
* Pregnant women
* body weight > 120 kg
* Neurological disease
* Fibromyalgia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Disability | Baseline, week 4 (end of intervention period)
  The change of the Oswestry Disability Index (ODI) between baseline and the end of the intervention period (4 weeks)

SECONDARY OUTCOMES:
Disability | week2 (intervention period); month 1, month 3 and month 6 follow-up period
  The change in the ODI score between baseline and follow-up period
Disability responding rate | week 2, week 4 (intervention period) and at month 1, month 3 and month 6 follow-up period
  Number and percentage of patients presenting an improvement from baseline of at least 10 points in the ODI
Back Pain | week 1, week 2, week 3 and week 4 (the intervention period)
  Changes in the average back pain intensity over the last week from baseline, assessed on Numerical Pain Rating Scale from 0 to 10 (0 for no pain and 10 for worst pain imaginable)
Back Pain | month 1, month 3 and month 6 (follow-up period)
  Changes in average back pain intensity over the last week from end of the intervention period (week 4), assessed on Numerical Rating Scale from 0 to 10 (0 for no pain and 10 for worst pain imaginable) in the follow-up period.
Back Pain responding rate | week 2, week 4 (intervention period) and at month 1, month 3 and month 6 (follow-up period)
  Number and percentage of patients presenting an improvement from baseline of at least 1.5 points in the Numerical Pain rating scale
Function | week 4
  Change in function score from baseline, assessed using the Pain Specific Functional Scale. The PSFS requires participants to identify three problematic activities and to rate these activities on a scale from 0 to 10.
Function | Between end of intervention period and month 1, month 3 and 6 post-intervention
  Change in function score from the end of the intervention period (week 4) in the follow-up period, assessed using the Pain Specific Functional Scale. The PSFS requires participants to identify three problematic activities and to rate these activities on a scale from 0 to 10.
Function responding rate | week 4 (intervention period) and at month 1, month 3 and month 6 (follow-up period)
  Number and percentage of patients presenting an improvement of at least 1.5 points from baseline in the pain specific function scale
Kinesiophobia | week 4
  Change in fear of movements and attitudes and behavior from baseline towards pain score, evaluated through the Tampa questionnaire.
Kinesiophobia | month 1, month 3 and 6 (follow-up period)
  Change in fear of movements and attitudes and behavior from the end of intervention period (week4), towards pain score, evaluated through the Tampa questionnaire.
Kinesiophobia responding rate | week 4 (intervention period) and month 1, month 3 and month 6 (follow-up period)
  Number and percentage of patients presenting an improvement of at least 6 points from baseline in Tampa scale.
Anxiety and depression | week 4
  Change in Anxiety and depression score from baseline, assessed by the HAD questionnaire
Anxiety and depression | month 1, month 3 and 6 (follow-up period)
  Change in Anxiety and depression score from end of the intervention period (week 4), assessed by the HAD questionnaire.
Anxiety and depression responding rate | week 4 (intervention period) and month 1, month 3 and month 6 (follow-up period)
  Number and percentage of patients presenting an improvement of at least 2 points from baseline for each sub-scale anxiety and depression in the two treatment arms
Physiotherapist global satisfaction | week 4
  A single score of satisfaction reported by the physiotherapist:
  * How satisfied or dissatisfied are you with the ability of the LumbaCure® intervention to improve your patient low back pain condition (7-points scale; 1 = completely dissatisfied; 7 = completely satisfied); ?
  * How satisfied or dissatisfied are you with the ability of the Physical exercises intervention to improve your patient low back pain condition (7-points scale; 1 = completely dissatisfied; 7 = completely satisfied)?
Patient global satisfaction of the therapy | End of intervention period (week 4)
  A single score of satisfaction will be calculated based on a set of two questions:
  > How satisfied or dissatisfied are you with the ability of the LumbaCure® / Physical exercises intervention to improve your low back pain condition (7-points scale; 1 = completely dissatisfied; 7 = completely satisfied)? How globally would you rate your experience, on the LumbaCure® device/with physical exercises (7-point Likert scale (1 = very bad; 7 = excellent)) ?

OTHER OUTCOMES:
Patient mobilization | LumbaCure® session 1 and session 12 : Week 1 (Day 0) and Week 4 (Day 25)
  o Pressure distribution using a pressure mat
Measurement in Dynamic/static situation | Baseline and week 4 (end of intervention period)
  During standardized everyday dynamic/static movements (5x) : "sit-to-stand", 5 repetitions; climbing stairs", 5 repetitions; and "bending task", 30 sec position maintenance:
  - Patient muscular activation of the back muscles is measured by surface EMG (sEMG). Targeted muscles: Iliocostalis, longissimus, multifidus, obliques.
Measurement in Dynamic/static situation | Baseline and week 4 (end of intervention period)
  During standardized everyday dynamic/static movements (5x) : "sit-to-stand", 5 repetitions; climbing stairs", 5 repetitions; and "bending task", 30 sec position maintenance:
  - Patient Trunk acceleration, measured by IMU.
Flexion/extension amplitudes | Baseline and week 4 (end of intervention period)
  Flexion/extension amplitudes measured using the Tergumed or DavidBack device.
Force | Baseline and week 4 (end of intervention period)
  Force measured using the Tergumed or DavidBack device.
Distance finger to floor | Baseline and week 4 (end of intervention period)
  The ability of the patient to flex the lower back via fingertips to floor distance.
Adverse events | baseline, week 1, week 2, week 3, week 4
  The occurrence, intensity and severity of adverse events will be monitored on both arm

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Jessa Ziekenhuis vzw, Hasselt
  - Jessa Ziekenhuis vzw, Herk-de-Stad

IPD SHARING:
Plan to Share IPD: No